CLINICAL TRIAL: NCT07172477
Title: Early Feasibility Study (EFS) of the 'Pivot Extend' for the Treatment of Tricuspid Regurgitation, Including High-Risk Patients (SPACER Study, Australia)
Brief Title: Early Phase Study Using the 'Pivot Extend' System as a Treatment for Patients With Tricuspid Regurgitation
Acronym: SPACER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tau Medical Australia Pty Ltd (Industry)
Collaborators: Tau-MEDICAL Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Tau-MEDICAL Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCP-EFS-12-AU
Record Dates: First submitted 2025-08-19; First posted 2025-09-15 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Tricuspid Regurgitation
Keywords: Tricuspid Regurgitation; SPACER; Pivot Extend
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pivot Extend device (Experimental): Patients aged 18 years or older with severe and symptomatic tricuspid regurgitation
  Interventions: Device: Pivot Extend

INTERVENTIONS:
Device: Pivot Extend — The investigational "Pivot Extend" device will be inserted through a small incision in the femoral vein and guided to the heart using a catheter. The Pivot Extend device is designed to sit in the space where the valve isn't closing, helping the flaps of the valve to close tightly and reducing the amount of blood leaking back through the valve.

SUMMARY:
Participants with severe tricuspid regurgitation may require heart surgery to repair or replace the tricuspid valve. However, there is a high risk associated with these surgeries and it is often not feasible for elderly patients or those with other medical conditions.

The goal of this clinical investigation is

* To assess the safety of the investigational device "Pivot Extend" in participants aged 18 years or over with severe and clinically symptomatic Tricuspid Regurgitation (TR) deemed suitable for percutaneous valve intervention
* To evaluate device success, procedural success and clinical outcomes in improving TR symptoms following implantation of the "Pivot Extend" device

ELIGIBILITY:
Inclusion Criteria:

* Has voluntarily decided to participate in this clinical trial and has provided written informed consent
* Adults aged 18 years or older at the time of informed consent
* Has symptoms of TR corresponding to at least NYHA Class II, despite receiving optimal medical therapy for at least 30 days prior to screening
* Meets the criteria at least severe (3+) on the TR grade classification table on echocardiography performed at the screening visit
* Deemed suitable for percutaneous valve intervention by a Heart Team that includes at least one cardiologist and one cardiac surgeon
* Is able to understand and follow the investigator's instructions and is able to participate for the entire duration of the study

Exclusion Criteria:

* Has blood clots, emboli, masses, or growths in the vascular system of the heart or lungs on an echocardiogram and cardiac CT scan performed at the screening visit
* Uncorrected blood clotting disorders based on hematology tests performed at the screening visit
* Unable to use anticoagulant agents (NOAC ex.Xarelto)
* A history of major bleeding (excluding minor bleeding such as nosebleed that can be hemostasized) treated with anticoagulants at any time prior to participation in this clinical trial
* Severe anemia (hemoglobin less than or equal to 80g/L)
* Has an implanted device such as an implantable cardioverter defibrillator (ICD) or pacemaker
* Has anatomy that, in the opinion of the investigator, is not suitable for implantation of an investigational medical device based on echocardiogram and cardiac CT scan performed at the screening visit
* Requires surgery or interventional procedures (coronary artery bypass graft (CABG) or surgery for atrial septal defect (ASD)) based on an echocardiogram performed at the screening visit
* Platelet count of 50 x 10^9 per litre of blood or less based on hematology tests performed at the screening visit
* Pulmonary arterial hypertension, defined as pulmonary artery systolic pressure greater than 70mmHg on cardiac catheterization performed at the screening visit, or a pulmonary vascular resistance greater than 3 Wood Units on right heart catheterization
* Left ventricular ejection fraction (LVEF) of less than 20% on echocardiogram performed at the screening visit
* Active gastrointestinal bleeding or a digestive procedure within 90 days prior to screening for this study, and/or those with the potential for gastrointestinal bleeding in the opinion of the investigator
* History of cerebrovascular accident (CVA) or transient ischemic attacks (TIA) within 30 days prior to screening for this clinical trial
* History of myocardial infarction (MI) within 30 days prior to screening for this study
* Active endocarditis requiring antibiotic treatment
* Malignancies or end-stage renal failure requiring hemodialysis and other chronic conditions with a life expectancy of less than one year
* Moderate or severe aortic, pulmonary artery, or mitral stenosis on echocardiogram performed at the screening visit
* Severe or greater mitral valve regurgitation or severe aortic valve regurgitation as determined by echocardiographic grading criteria at the screening visit
* Calcification of the tricuspid valve leaflets affecting the procedure on an echocardiogram performed at the screening visit
* Those who have participated in another clinical trial within 30 days prior to screening for this clinical trial
* Pregnant or breastfeeding, or planning to become pregnant during the clinical trial period
* Participants of childbearing potential who are not using a highly effective method of contraception
* Coexisting condition, which most likely limits the life expectancy to less than one year
* Preexisting pulmonary valve prosthesis or a right ventricle to pulmonary artery (RV-PA) conduit
* Any other clinical findings that, in the opinion of the investigator, are medically inappropriate for this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of the implantation of the "Pivot Extend" device | 30 days post device implantation
  Occurrence rate of major adverse cardiac events (MACE) (e.g. stroke, myocardial infarction, pulmonary embolism)

SECONDARY OUTCOMES:
To evaluate the Pivot Extend device success | During implantation procedure
  Rate of successful device placement at target location
To evaluate the procedural success (1) | 30 days, 180 days and 365 days post device implantation
  The number of participants who experienced at least 1 drop in their TR grade from screening, based on echocardiographic assessment
To evaluate the procedural success (2) | 30 days, 180 days and 365 days post device implantation
  Changes in echocardiogram (measurements and assessments of the heart's structure and function) as assessed by the central "Core Lab" reader
To evaluate the procedural success (3) | 180 and 365 days after device implantation
  Occurrence rate of MACE associated with the device or procedure
To evaluate the procedural success (4) | 30 days, 180 days and 365 days post device implantation
  Changes in Computed Tomography (CT) images (evaluating the size, shape and function of the tricuspid valve following Pivot Extend device insertion) as assessed by the central "Core Lab" reader.
To evaluate the clinical outcomes (1) | 180 days and 365 days post device implantation
  Changes in right ventricular volume from baseline, assessed by cardiac computed tomography (CT)
To evaluate the clinical outcomes (2) | 180 days and 365 days post device implantation
  Changes in echocardiogram (measurements and assessments of the heart's structure and function) as assessed by the central "Core Lab" reader
To evaluate the clinical outcomes (3) | 30 days, 180 days and 365 days post device implantation
  Number of participants with improvement in New York Heart Association (NYHA) functional class (system to classify the severity of heart failure symptoms) from baseline
To evaluate clinical outcomes (4) | 30 days, 180 days and 365 days post device implantation
  Measure in the changes of distance travelled during a 6 Minute Walk Test from baseline
To evaluate clinical outcomes (5) | 30 days, 180 days and 365 days post device implantation
  Changes in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) score (a measure of symptoms, physical limitation, social limitations and quality of life domains) from baseline. Participants will be asked to tick a box on a scale indicating how each domain affects their life (e.g. scales range from extremely limited to not at all limited, from every morning/night to never over the past 2 weeks, from completely dissatisfied to completely satisfied). The responses will be used to calculate an average score on a scale of 0 to 100. A higher score equates to better outcomes (i.e. fewer symptoms, better physical and social function, improved quality of life).
To evaluate clinical outcomes (6) | 30 days, 180 days and 365 days post device implantation
  Number of participants with at least 1 level of improvement in pitting edema from baseline
To evaluate clinical outcome measures (7) | 30 days, 180 days and 365 days post device implantation
  Changes in eGFR (estimated glomerular filtration rate) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: June-Hong Kim, PhD, Study Director — Tau-MEDICAL Co., Ltd.
Locations (1):
- Macquarie University, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No